CLINICAL TRIAL: NCT00002911
Title: A PHASE III, MULTI-CENTER, RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED STUDY OF MARIMASTAT IN PATIENTS WITH MINIMAL DISEASE STAGE III NON-SMALL CELL LUNG CANCER
Brief Title: Marimastat in Treating Patients With Stage III Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ILEX Oncology Services, Incorporated (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000065284; ILEX-C03-IVB/173; BB-C03-IVB/173; NCI-V96-1113
Record Dates: First submitted 1999-11-01; First posted 2004-05-26 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2007-05

CONDITIONS: Lung Cancer
Keywords: stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — marimastat

INTERVENTIONS:
Drug: marimastat

SUMMARY:
RATIONALE: Marimastat may stop the growth of non-small cell lung cancer by stopping blood flow to the tumor.

PURPOSE: Randomized double-blinded phase III trial to determine the effectiveness of marimastat in treating patients who have residual stage III non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the effect of marimastat (a matrix metalloproteinase inhibitor) vs. placebo on overall survival in patients with Stage III non-small cell lung cancer who have minimal residual disease following chemotherapy, radiotherapy, and/or surgery. II. Assess the effect of marimastat on time to disease progression in these patients. III. Assess the safety and tolerability of marimastat in these patients.

OUTLINE: This is a randomized, double-blind study. Patients are randomized no less than 2 and no more than 8 weeks after the last prior treatment modality received. Patients are stratified by participating institution. Patients are randomly assigned to receive either oral marimastat or oral placebo twice daily. Treatment begins within 5 days of minimization and continues for up to 18 months after the last patient is enrolled, unless disease progression or unacceptable toxicity intervenes. Patients deriving benefit at end of study may continue treatment if desired. Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 504 patients will be entered over 30 months from approximately 60 centers.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed non-small cell lung cancer Stage IIIA/B disease No malignant pleural effusions Minimal residual disease after one or a combination of the following: Incomplete surgical resection i.e., macroscopic residual disease at completion of surgery Radical radiotherapy with no evidence of disease progression at entry Documented complete or partial tumor response following at least 2 courses of cytotoxic chemotherapy No evidence of disease progression during or following prior therapy

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Hematopoietic: Absolute neutrophil count greater than 500/mm3 Platelet count greater than 50,000/mm3 Hepatic: Bilirubin less than 2.0 times upper limit of normal (ULN) AST/ALT no greater than 3.0 times ULN Renal: Creatinine no greater than 1.5 times ULN Other: No acute illness within 1 week of start of study No other illness that would significantly interfere with study outcome No major medical illness that precludes prolonged marimastat administration No second malignancy within 5 years except: Adequately treated basal cell carcinoma of the skin In situ carcinoma of the cervix Not pregnant or nursing Medically approved method of contraception required of fertile women Willing and able to tolerate and comply with study requirements

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: See Disease Characteristics No prior marimastat, batimastat, bleomycin, or busulphan No more than 1 cytotoxic chemotherapy regimen for non-small cell lung cancer Endocrine therapy: Not specified Radiotherapy: See Disease Characteristics Surgery: See Disease Characteristics Other: At least 4 weeks since any investigational drug therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1996-12; Study Completion 2004-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Heck, MEd, MBA, Study Chair — ILEX Oncology Services, Incorporated
Locations (50):
- United States (48):
  - Comprehensive Cancer Institute of Huntsville, Huntsville, Alabama
  - Hematology Associates, Ltd., Phoenix, Arizona
  - Marin Cancer Institute, Greenbrae, California
  - Scripps Clinic, La Jolla, California
  - Scripps Memorial Hospital Stevens Cancer Center, La Jolla, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - St. Joseph Hospital - Orange, Orange, California
  - John Wayne Cancer Institute, Santa Monica, California
  - Kaiser Permanente Medical Center - Vallejo, Vallejo, California
  - Rocky Mountain Cancer Center, Denver, Colorado
  - University of Colorado Cancer Center, Denver, Colorado
  - University of Connecticut Health Center, Farmington, Connecticut
  - Vincent T. Lombardi Cancer Research Center, Georgetown University, Washington D.C., District of Columbia
  - Comprehensive Cancer Center at JFK Medical Center, Atlantis, Florida
  - Radiation Therapy Associates - Fort Myers, Fort Myers, Florida
  - Oncology-Hematology Group of South Florida, Miami, Florida
  - Bay Area Oncology, MD'S, PA, Tampa, Florida
  - Rush-Presbyterian-St. Luke's Medical Center, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Community Hospitals of Indianapolis - Regional Cancer Center, Indianapolis, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Veterans Affairs Medical Center - Lexington, Lexington, Kentucky
  - Louisiana State University School of Medicine, New Orleans, Louisiana
  - Hubert H. Humphrey Cancer Center, Coon Rapids, Minnesota
  - St. Louis University Health Sciences Center, St Louis, Missouri
  - Southwest Cancer Clinic, Henderson, Nevada
  - Cancer Institute of New Jersey at Hamilton, Hamilton, New Jersey
  - Beth Israel Medical Center, New York, New York
  - Kaplan Cancer Center, New York, New York
  - Strong Memorial Hospital of the University of Rochester, Rochester, New York
  - Barrett Cancer Center, The University Hospital, Cincinnati, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - Natalie Warren Bryant Cancer Center, Tulsa, Oklahoma
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Hematology-Oncology Mawr Medical North, Bryn Mawr, Pennsylvania
  - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Care Group, Philadelphia, Pennsylvania
  - Allegheny University Hospitals - Graduate MCP, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Pittsburgh Pediatric Research, Inc., Pittsburgh, Pennsylvania
  - Roger Williams Medical Center/BUSM, Providence, Rhode Island
  - Jackson Clinic Professional Association, Jackson, Tennessee
  - Baptist Regional Cancer Center - Knoxville, Knoxville, Tennessee
  - Texas Oncology PA (TOPA) at Baylor-Sammons, Dallas, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Joe Arrington Cancer Research and Treatment Center, Lubbock, Texas
- Canada (2):
  - Ottawa Regional Cancer Center - General Division, Ottawa, Ontario
  - Toronto General Hospital, Toronto, Ontario